CLINICAL TRIAL: NCT01264276
Title: Telemedicine Approaches to Evaluating Acute-phase ROP
Acronym: e-ROP
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Johns Hopkins University (Other); Boston Children's Hospital (Other); Nationwide Children's Hospital (Other); Duke University (Other); University of Louisville (Other); University of Minnesota (Other); University of Oklahoma (Other); The University of Texas at San Antonio (Other); University of Utah (Other); University of Pennsylvania (Other); Vanderbilt University (Other); University of Calgary (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10-007554; U10EY017014-01A2 (NIH)
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Retinopathy of Prematurity
Keywords: ROP; Retinopathy of Prematurity; Telemedicine
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary objective of this multi-center clinical study is to evaluate the validity, reliability, feasibility, safety and relative cost-effectiveness of a retinopathy of prematurity (ROP) telemedicine evaluation system to detect eyes of at-risk babies who meet referral warranted ROP (RW-ROP) criteria and therefore need a diagnostic evaluation by an ophthalmologist experienced in ROP.

We shall:

1. Calculate the accuracy, using sensitivity and specificity, of the system to provide remote evaluations when compared with the findings of a "gold standard" indirect ophthalmoscopic examination performed by a Study-certified ophthalmologist, rigorously trained in ROP diagnostic examinations (validity);
2. Determine intra-reader and inter-reader agreement for deciding whether digital images indicate that the eyes of a baby are in need of diagnostic indirect ophthalmoscopy by an ophthalmologist experienced in ROP (reliability);
3. Determine whether imaging evaluation can be achieved for each baby (feasibility);
4. Examine ocular and systemic complications associated with digital imaging and compared with those associated with diagnostic examinations performed by an ophthalmologist (safety);
5. Compare the costs and benefits of adopting a telemedicine retinal imaging system compared to the current cost of indirect ophthalmoscopic examinations (cost-effectiveness).

DETAILED DESCRIPTION:
Eligibility Criteria:

• Babies with birth weights of <1251 grams(g) at selected large clinical centers in the US and Canada.

Procedures:

• Participants will undergo both digital retinal imaging and clinically indicated indirect ophthalmoscopic examinations on the same day. Wide-field digital images (WF-DI) of both eyes will be captured by non-physician Certified ROP Imagers (CRIs) using standardized imaging protocols. The RetCam Shuttle® (Clarity Medical Systems, Pleasanton, CA), a corneal-contact camera that captures wide field (130 degree field of view) retinal images, will be used.

Masking:

• Study-certified Ophthalmologist and Study-certified Imager at the clinical sites will be masked to each other's findings. The Study Clinical Coordinator (SCC) will remain unmasked. SCC will monitor the clinical noteworthy events and report all adverse events to the site Institutional Review Board (IRB), the Project Director at the Office of Study Chair, and to the Data Coordinating Center (DCC). DCC will prepare closed-session Data Monitoring and Oversight Committee (DMOC) reports. The PI at each site will monitor adverse events.

Outcome Measures:

• The primary outcome measure is detection of referral warranted ROP (RW-ROP) on digital images. Retinal images will be graded by Trained Readers using a standardized protocol to identify eyes with RW-ROP. Results of the gradings will be compared to the diagnostic examinations being performed on each child at the same session when images taken. For comparison, images will also be graded by ROP experts (Expert Readers).

ELIGIBILITY:
Inclusion Criteria:

* Babies with birth weighs of <1251g at selected large clinical centers in the US and Canada.
* Admitted to a participating Neonatal Intensive Care Units (NICU) and expected to survive to 28 days.
* Likely to remain in participating NICU for serial ROP exams.
* Transferred to participating NICU for treatment of ROP (regardless of PMA).
* Parents or guardians have provided informed consent for participation in the study.

Exclusion Criteria:

* Failure to obtain informed consent.
* Known ocular anomalies that prevent imaging of the retina.
* Life threatening anomalies (i.e. heart, neurological, etc).
* Admission to participating NICU with ROP that is already regressing or treated.

Ages: 32 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Babies with birth weighs of <1251g at selected large clinical centers in the US
Sampling Method: Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2011-07; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Detection of Referral Warranted ROP | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Graham E Quinn, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (12):
- United States (11):
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Duke University, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Wade KC, Ying GS, Baumritter A, Gong A, Kemper AR, Quinn GE; e-ROP Cooperative Group. Factors in Premature Infants Associated With Low Risk of Developing Retinopathy of Prematurity. JAMA Ophthalmol. 2019 Feb 1;137(2):160-166. doi: 10.1001/jamaophthalmol.2018.5520. PMID 30452500
- [Derived] Morrison D, Bothun ED, Ying GS, Daniel E, Baumritter A, Quinn G; e-ROP Cooperative Group. Impact of number and quality of retinal images in a telemedicine screening program for ROP: results from the e-ROP study. J AAPOS. 2016 Dec;20(6):481-485. doi: 10.1016/j.jaapos.2016.08.004. Epub 2016 Oct 1. PMID 27702612
- [Derived] Quinn GE, Ying GS, Repka MX, Siatkowski RM, Hoffman R, Mills MD, Morrison D, Daniel E, Baumritter A, Hildebrand PL, Schron EB, Ells AL, Wade K, Kemper AR. Timely implementation of a retinopathy of prematurity telemedicine system. J AAPOS. 2016 Oct;20(5):425-430.e1. doi: 10.1016/j.jaapos.2016.06.007. Epub 2016 Sep 17. PMID 27651231
- [Derived] Kemper AR, Prosser LA, Wade KC, Repka MX, Ying GS, Baumritter A, Quinn GE; e-ROP Study Cooperative Group. A Comparison of Strategies for Retinopathy of Prematurity Detection. Pediatrics. 2016 Jan;137(1):e20152256. doi: 10.1542/peds.2015-2256. Epub 2015 Dec 15. PMID 26672022
- [Derived] Wade KC, Pistilli M, Baumritter A, Karp K, Gong A, Kemper AR, Ying GS, Quinn G; e-Retinopathy of Prematurity Study Cooperative Group. Safety of Retinopathy of Prematurity Examination and Imaging in Premature Infants. J Pediatr. 2015 Nov;167(5):994-1000.e2. doi: 10.1016/j.jpeds.2015.07.050. Epub 2015 Aug 20. PMID 26299381
- [Derived] Kemper AR, Wade KC, Hornik CP, Ying GS, Baumritter A, Quinn GE; Telemedicine Approaches to Evaluating Acute-phase Retinopathy of Prematurity (e-ROP) Study Cooperative Group. Retinopathy of prematurity risk prediction for infants with birth weight less than 1251 grams. J Pediatr. 2015 Feb;166(2):257-61.e2. doi: 10.1016/j.jpeds.2014.09.069. Epub 2014 Nov 12. PMID 25449219
- [Derived] Quinn GE, Ying GS, Daniel E, Hildebrand PL, Ells A, Baumritter A, Kemper AR, Schron EB, Wade K; e-ROP Cooperative Group. Validity of a telemedicine system for the evaluation of acute-phase retinopathy of prematurity. JAMA Ophthalmol. 2014 Oct;132(10):1178-84. doi: 10.1001/jamaophthalmol.2014.1604. PMID 24970095
- [Derived] Graham E Quinn; e-ROP Cooperative Group. Telemedicine approaches to evaluating acute-phase retinopathy of prematurity: study design. Ophthalmic Epidemiol. 2014 Aug;21(4):256-67. doi: 10.3109/09286586.2014.926940. Epub 2014 Jun 23. PMID 24955738